CLINICAL TRIAL: NCT06841367
Title: The Effect of Awareness-Based Stress Reduction Training on Anxiety Level and Physiological Parameters in Pregnant Women Diagnosed With Preeclampsia
Brief Title: The Effect of Awareness-Based Stress Reduction Training on Preeclampsia and Anxiety
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, SERTAP MANTARCI, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011-KAEK-55
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Preeclampsia Mild to Moderate
Keywords: preeclampsia; anxiety level; physiological parameters
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Intervention Model Description: It is a study with a randomized controlled experimental design. Two groups with preeclampsia will be included in the study. Experimental group (group receiving mindfulness training), Control group (group without intervention)
Who Masked: Participant
Masking Description: The control group will not receive mindfulness-based stress reduction training, and outcome assessments will be conducted by a researcher dependent on group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mindfulness-based stress reduction training (Experimental): The participants' anxiety levels and physiological parameters will be measured at the initial stage. For 8 weeks in the intervention group, conscious awareness-based stress reduction training will be given online for 1 hour a week. Control at week 4 and Interim evaluations will be provided for intervention groups. At the end of the 8th week, anxiety level and physiological parameters were again will be evaluated.
  Interventions: Other: Mindfulness-based stress reduction training
- Control group (No Intervention): The participants' anxiety levels and physiological parameters will be measured at the initial stage. No intervention will be made to the control group. Physiological parameters and anxiety levels will be measured at the 4th and 8th weeks.

INTERVENTIONS:
Other: Mindfulness-based stress reduction training — It is expected that improvements in physiological parameters and anxiety levels will be observed in the preeclampsia group with awareness-based stress reduction training.
  Arms: mindfulness-based stress reduction training

SUMMARY:
Preeclampsia is a multisystem disease that occurs during pregnancy and carries risks into the postpartum period. This condition, which threatens maternal and fetal health, requires close monitoring and good care. Pregnant women need to rely on both their previously used coping mechanisms and learn new coping methods to manage the stress associated with high-risk pregnancies. Complementary and integrative therapies are utilized in managing hypertensive disorders and anxiety during pregnancy. Literature reviews show that complementary medicine practices included in current care may be effective in alleviating the symptoms of preeclampsia and reducing anxiety levels. However, the existing scientific studies are not at a sufficient level of evidence, and more advanced studies are needed in this area.

The aim of our thesis study is to examine the effect of mindfulness-based stress reduction training on anxiety levels and physiological parameters in pregnant women diagnosed with preeclampsia.

DETAILED DESCRIPTION:
Preeclampsia is a condition characterized by hypertension and proteinuria that occurs after the 20th week of pregnancy. The anxiety and fear experienced by pregnant women diagnosed with preeclampsia about their own and their baby's well-being lead to an increase in anxiety levels.

Mindfulness has been defined as the awareness of one's present-moment experience, accompanied by an attitude of kindness, friendliness, and non-judgmental acceptance .

Mindfulness-Based Stress Reduction (MBSR) is a clinical program that provides systematic training in mindfulness meditation as a self-regulation approach to facilitate adjustment to medical conditions, reduce stress, and manage emotions.

In a study conducted to determine the effect of mindfulness training on lowering blood pressure in preeclamptic women, a decrease in systolic and diastolic blood pressure was observed.

A study examining the effects of mindfulness training on maternal anxiety and self-efficacy in relation to childbirth found that anxiety levels decreased in pregnant women, and it was recommended that healthcare providers and pregnant women participate in mindfulness programs to improve pregnancy outcomes and childbirth.

It has been determined that mindfulness-based interventions during pregnancy can be beneficial for outcomes such as anxiety, depression, perceived stress, and mindfulness levels in the perinatal period.

Mindfulness-based training for the psychological health of pregnant women has been reported to significantly reduce perceived stress and depression, while increasing mindfulness and self-efficacy in women.

Mindfulness-based stress reduction training aimed at examining its effects on stress, anxiety, and prenatal attachment in high-risk pregnancies was found to reduce anxiety, increase prenatal attachment, and have no effect on stress levels in pregnant women .

A meta-analysis examining the effects of diet, exercise, yoga, and mindfulness practices during pregnancy to prevent hypertensive disorders found that these lifestyle interventions reduced the incidence of hypertension in pregnancy.

The aim of our thesis study is to examine the effect of mindfulness-based stress reduction training on anxiety levels and physiological parameters in pregnant women diagnosed with preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Knowing Turkish
* Being literate
* Being over 18
* Being primiparous
* Having a singleton fetus and cephalic presentation
* Being diagnosed with preeclampsia
* Agreeing to participate in the study

Exclusion Criteria:

* Having any additional disease other than preeclampsia
* Participant's voluntary withdrawal from the study
* Having a cesarean section for any reason

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — It is aimed to ensure that pregnant women are minimally affected by the preeclampsia diagnosis they receive.
Enrollment: 80 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-05-05 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory | two months
  The State-Trait Anxiety Inventory was developed by Spielberger and colleagues to measure state anxiety and trait anxiety. The final value obtained represents the individual's anxiety score. The scores obtained from both scales theoretically range between 20 and 80. A higher score indicates a higher level of anxiety. A lower score indicates a lower level of anxiety.

SECONDARY OUTCOMES:
measurement of physiological parameters / arterial blood | two months
  Arterial blood pressure will be measured with a manual device and a stethoscope. Blood pressure will be expressed in mmHg. Blood pressure values above 140/90 mmHg will be considered high, while values below 140/90 mmHg will be considered normal.
measurement of physiological parameters / heart rate | two months
  The heart rate will be measured by counting the brachial artery beats for 60 seconds with the help of a stopwatch. The unit will be expressed as beats per minute (bpm).
measurement of physiological parameters / fever | two months
  Fever will be measured with a thermometer. The unit for the fever parameter is expressed in °C. Fever values below 36.0 °C and above 37.5 °C will be considered abnormal.

CONTACTS AND LOCATIONS:
Overall Officials: Istanbul University-Cerrahpaşa Faculty of Health Sciences Postgraduate Education Institute, ASSOCIATE PROFESSOR, Principal Investigator — husniye.dinckaya@iuc.edu.tr; SERTAP MANTARCI, MIDWIFERY GRADUATE STUDENT, Principal Investigator — sertap.mantarci@gmail.com

IPD SHARING:
Plan to Share IPD: No